CLINICAL TRIAL: NCT03172884
Title: An Open-label Non-randomized, Phase 1 Single Dose Study to Evaluate the Pharmacokinetics and Safety of Copanlisib in Subjects With Impaired Hepatic or Renal Function in Comparison to Healthy Subjects
Brief Title: Study of Copanlisib in Hepatic or Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18041; 2016-004561-51 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hepatic Insufficiency, Renal Insufficiency
Keywords: Renal Impairment; Pharmacokinetics; Hepatic impairment; Envisaged indication: Treatment of cancer
MeSH Terms: conditions — Hepatic Insufficiency; Renal Insufficiency | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAY80-6946/Healthy subject (Experimental): Healthy subjects
  Interventions: Drug: Copanlisib (ALIQOPA, BAY80-6946)
- BAY80-6946/moderate hepatically impaired patients (Experimental): Patients with Child-Pugh B (score 7-9) at the screening visit
  Interventions: Drug: Copanlisib (ALIQOPA, BAY80-6946)
- BAY80-6946/severe renal impaired patients (Experimental): Patients with eGFR 15-29 mL/min/1.73 m^2 at the screening visit based on the Modification of Diet in Renal Disease (MDRD) equation
  Interventions: Drug: Copanlisib (ALIQOPA, BAY80-6946)
- BAY80-6946/severe hepatically impaired patients (Experimental): Patients with Child-Pugh C (score 10-15) at the screening visit
  Interventions: Drug: Copanlisib (ALIQOPA, BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (ALIQOPA, BAY80-6946) — 12mg single dose, intravenous on Day 0

SUMMARY:
To evaluate the pharmacokinetics and safety of copanlisib in subjects with impaired hepatic or renal function in comparison to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

All subjects - Male and female subjects between 18 and 80 years of age with a body mass index above 18.0 and below 34.0 kg / m² and a body weight of above or equal 50 kg.

Healthy subjects

- Healthy subjects as determined by absence of clinically significant deviation from normal in medical history, physical examination, vital signs, electrocardiograms, and clinical laboratory determinations. eGFR ≥ 90 mL/min/1.73 m² (according to Modification of Diet in Renal Disease [MDRD] formula).

Subjects with moderate or severe hepatic impairment

* Subjects with confirmed liver cirrhosis by at least one of the following Criteria: histologically by prior liver biopsy showing cirrhosis, liver imaging (computer tomography, and/or ultrasound and/or magnetic resonance imaging scans, and/or fibroscan), or laparoscopy.
* Child-Pugh Clinical Assessment Score 7 to 9 (moderate) or Score 10 to 15 (severe).

Subjects with severe renal impairment

* Subjects with severe renal impairment with an estimated glomerular filtration rate 15-29 mL/min/1.73 m² according to MDRD formula.
* Subjects with stable renal disease: no significant change in renal function as evidenced by serum creatinine value within ±25% from the last determination, obtained within at least 3 months before study entry and the absence of the need to start dialysis in the next 3 months.

Exclusion Criteria:

All subjects

* Active coronary artery disease or myocardial infarction within 6 months of study entry. Immuno-compromised subjects including known history/seropositivity of human immunodeficiency virus (HIV).
* Other concurrent severe and/or uncontrolled medical conditions (e.g. current diagnosis of type 1 or type 2 diabetes mellitus and with HbA1c >8.5%) that could cause unacceptable safety risks or compromise compliance with protocol.
* Previous or concurrent history of malignancies within 5 years prior to study treatment except for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder cancer as well as localized prostate cancer.
* Uncontrolled hypertension despite optimal medical management (per investigator's assessment).
* Administration of strong CYP3A4 inhibitors or inducers within 2 weeks prior to dosing and during study conduct. (A list of these medications can be found in Section 16.6 of the protocol. However, this list may not be comprehensive).

Subjects with moderate or severe hepatic impairment

* Symptoms or history of encephalopathy (Grade III or worse)
* Failure of any other major organ other than the liver; severe infection, or any clinically significant illness within 4 weeks prior to study drug administration
* Renal failure with an eGFR <35 mL/min/1.73 m² Subjects with severe renal impairment
* Acute renal failure at study entry
* Nephrotic syndrome
* Failure of any other major organ other than the kidney
* Acute hepatorenal syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany
- Institutul National de Boli Infectioase Prof.Dr.Matei Bals, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, time point and process of data access. As such, Bayer commits to sharing upon request from qualified researcher's patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in Germany and Romania between 14 Jun 2017 (first patient's first visit) and 13 Mar 2020 (last patient's last visit).
Pre-assignment Details: 50 participants were screened in study. 16 were screen failure and 4 withdrew from study. 30 participants were assigned to study arms.
Groups:
- Moderate Hepatic Impairment Group: Child-Pugh B (score 7-9) at the screening visit
- Severe Hepatic Impairment Group: Child-Pugh C (score 10-15) at the screening visit
- Severe Renal Impairment Group: eGFR 15-29 mL/min/1.73 m^2 at the screening visit based on the Modification of Diet in Renal Disease (MDRD) equation
- Healthy Participants: Normal hepatic and renal function group
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Started | 8 | 6 | 8 | 8
Completed | 8 | 6 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants | Total
Number analyzed (Participants) | 8 | 6 | 8 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.4) | 47.5 (11.1) | 65.8 (12.1) | 60.9 (6.6) | 60.7 (11.7)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 4 | 6 | 3 | 6 | 19
  From 65-84 years | 4 | 0 | 5 | 2 | 11
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 3 | 9
  Male | 5 | 5 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 8 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 6 | 8 | 8 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index: weight [kg] / (height [m])²
  kg/m^2 | 27.90 (4.68) | 27.12 (4.76) | 26.60 (3.07) | 26.48 (1.64) | 27.02 (3.53)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Copanlisib in Plasma.
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: before copanlisib administration as well as 10 min and 1 h (end of infusion), 1.5, 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120 and 168 h after start of infusion
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 6 | 8 | 8
μg/L | 68.12 (65.50) [lower limit 65.50] | 71.09 (53.90) [lower limit 53.90] | 31.77 (38.25) [lower limit 38.25] | 49.20 (27.24) [lower limit 27.24]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Participants; Moderate Hepatic Impairment vs Healthy Subjects; Test type: Other; LS means = 1.385, 90% CI 2-sided [0.921 to 2.081]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Healthy Participants; Severe hepatic impairment group vs Healthy Subjects; Test type: Other; LS means = 1.445, 90% CI 2-sided [0.998 to 2.093]
Statistical Analysis 3: Comparison: Severe Renal Impairment Group vs Healthy Participants; Severe renal impairment group vs Healthy Subjects; Test type: Other; LS means = 0.646, 90% CI 2-sided [0.486 to 0.858]

2. Primary Outcome: Area Under the Concentration vs. Time Curve From Zero to Infinity (AUC) of Copanlisib in Plasma.
Description: AUC refers to area under the concentration vs time curve from 0 to infinity which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 1
Population: Participants in PK population with available data are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 6 | 7 | 6
μg*h/L | 594.9 (53.85) | 940.7 (23.70) | 373.7 (59.08) | 347.8 (23.99)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Participants; Moderate Hepatic Impairment group vs Healthy Subjects; Test type: Other; LS Means = 1.711, 90% CI 2-sided [1.148 to 2.550]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Healthy Participants; Severe hepatic impairment group vs Healthy Subjects; Test type: Other; LS Means = 2.705, 90% CI 2-sided [2.115 to 3.460]
Statistical Analysis 3: Comparison: Severe Renal Impairment Group vs Healthy Participants; Severe renal impairment group vs Healthy Subjects; Test type: Other; LS Means = 1.075, 90% CI 2-sided [0.696 to 1.659]

3. Primary Outcome: Area Under the Concentration-time Curve of Copanlisib in Plasma Over the Time Interval From 0 to 168 h.
Description: AUC(0-168) refers to AUC from time 0 to 168 hr which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 6 | 8 | 8
μg*h/L | 551.4 (53.78) | 853.0 (26.39) | 350.5 (48.55) | 311.9 (23.55)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Participants; Moderate Hepatic Impairment group vs Healthy Subjects; Test type: Other; LS Means = 1.768, 90% CI 2-sided [1.251 to 2.498]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Healthy Participants; Severe hepatic impairment group vs Healthy Subjects; Test type: Other; LS Means = 2.735, 90% CI 2-sided [2.163 to 3.459]
Statistical Analysis 3: Comparison: Severe Renal Impairment Group vs Healthy Participants; Severe renal impairment group vs Healthy Subjects; Test type: Other; LS Means = 1.124, 90% CI 2-sided [0.815 to 1.549]

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Metabolite M-1.
Description: The morpholinone derivative M-1 is a minor copanlisib metabolite in plasma. The PK of metabolite M-1 is routinely analyzed in addition to the PK of the parent compound, although M-1 is not considered to be a major metabolite. Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 1
Population: Participants in PK population with available data are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 4 | 8 | 7
μg/L | 1.868 (53.16) | 1.356 (52.63) | 1.440 (50.36) | 1.543 (47.18)

5. Secondary Outcome: Area Under the Concentration-time Curve of Metabolite M-1 in Plasma Over the Time Interval From 0 to 168 h.
Description: The morpholinone derivative M-1 is a minor copanlisib metabolite in plasma. The PK of metabolite M-1 is routinely analyzed in addition to the PK of the parent compound, although M-1 is not considered to be a major metabolite. AUC from time 0 to 168h which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 1
Population: Participants in PK population with available data are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 4 | 8 | 7
μg*h/L | 82.62 (59.06) [lower limit 59.06] | 83.00 (35.34) [lower limit 35.34] | 67.12 (70.48) [lower limit 70.48] | 74.68 (76.75) [lower limit 76.75]

6. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events are considered to be treatment-emergent if they have started or worsened after first application of study medication up to 30 days after end of treatment with study medication.
Time Frame: Up to 30 days after end of treatment with study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 6 | 8 | 8
Participants
  Any Adverse events (AE's) | 0 | 0 | 2 | 2
  Any Serious adverse events (SAE's) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) in Different Severity.
Description: as for outcome 6
Time Frame: Up to 30 days after end of treatment with study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
Number analyzed (Participants) | 8 | 6 | 8 | 8
Participants
  Mild | 0 | 0 | 2 | 1
  Moderate | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first administration of study drug up to 30 days after end of treatment with study medication.
Groups:
- Moderate Hepatic Impairment Group: Subjects with Child-Pugh B (score 7-9) at the screening visit.
Arm/Group | Moderate Hepatic Impairment Group | Severe Hepatic Impairment Group | Severe Renal Impairment Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 2/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment Group (N=8) | Severe Hepatic Impairment Group (N=6) | Severe Renal Impairment Group (N=8) | Healthy Participants (N=8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center will refrain from making any publications and shall not publish any press releases or other public announcements or statements about this Agreement, the Study, the Results of the Study and/or the Study Drug without Bayer's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03172884/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03172884/SAP_001.pdf